CLINICAL TRIAL: NCT05237258
Title: Specialty Compared to Oncology Delivered Palliative Care for Patients With Acute Myeloid Leukemia
Acronym: SCOPE-L
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-646
Record Dates: First submitted 2022-02-02; First posted 2022-02-14 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Relapsed Adult AML; Primary Refractory Acute Myeloid Leukemia; High Risk Acute Myeloid Leukemia
Keywords: Relapsed Adult AML; Primary Refractory Acute Myeloid Leukemia; High Risk Acute Myeloid Leukemia; Caregivers
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Specialty Palliative Care (Experimental): - Participants will complete baseline self-report assessments at the time of informed consent
  Interventions: Behavioral: Specialty Palliative Care
- Primary Palliative Care (Experimental): - Participants will complete baseline self-report assessments at the time of informed consent
  Interventions: Behavioral: Primary Palliative Care

INTERVENTIONS:
Behavioral: Specialty Palliative Care — Participants assigned to specialty palliative care will be cared for by both oncology and palliative care clinicians during their hospital stays for AML.
  Arms: Specialty Palliative Care
Behavioral: Primary Palliative Care — Participants assigned primary palliative care will be cared for by oncology clinicians who have been trained in palliative care during the hospital stays for AML.
  Arms: Primary Palliative Care

SUMMARY:
This research study is evaluating whether primary palliative care is an alternative strategy to specialty palliative care for improving quality of life, symptoms, mood, coping, and end of life outcomes in patients with acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
Patients with newly diagnosed AML confront a sudden and life-threatening diagnosis, requiring an immediate disruption of their life and an urgent hospitalization to begin therapy. During their hospitalization for chemotherapy, patients with AML often experience difficult physical symptoms that negatively impact their quality of life and physical function. Patients with AML also experience significant psychological distress as they combat the abrupt onset of illness, uncertainty regarding their prognosis, physical and social isolation during hospitalization, and complete loss of independence. The abrupt onset of these symptoms can be distressing to both the patient and their family and friends (also called "caregivers").

Research has shown that early involvement of a team of clinicians specializing in lessening (or "palliating") these physical and emotional symptoms and helping patients and their caregivers cope with AML improves their quality of life and experience with their illness. This team is called "specialty palliative care" and consists of physicians and advanced practice providers who work closely and collaboratively with the oncology team to care for patients and caregivers. Research has also shown that training oncology clinicians to incorporate palliative care skills into their practice, called "primary palliative care," is an alternative strategy to having specialty palliative care clinicians care for patients with leukemia.

The purpose of this study is to determine whether specialty palliative care or primary palliative care is the best way to improve the quality of life and experience of patients with AML and their caregivers. This study will randomly assign hospitals to deliver either specialty palliative care or primary palliative care for patients with AML. Participants in this study will receive either specialty or primary palliative care during their hospital stays based upon which strategy their hospital has been assigned to. Participants assigned to specialty palliative care will be care for by both oncology and palliative care clinicians during their hospital stays for AML. Participants assigned to primary palliative care will be cared for by oncology clinicians who have been trained in palliative care during their hospital stays for AML.

ELIGIBILITY:
Inclusion Criteria:

* Patient Inclusion Criteria

  * Hospitalized patients (age ≥ 18 years) with high-risk AML defined as:
  * Patients with new diagnosis ≥ 60 years of age
  * An antecedent hematologic disorder
  * Therapy related-disease
  * Relapsed or primary refractory AML
  * Within five business days of initiating therapy with either a) intensive chemotherapy (7+3) or modification of this regimen on a clinical trial, or a similar intensive regimen requiring prolonged hospitalization; or b) hypomethylating agents +/- additional agents or modification of this regimen on a clinical trial.
* Caregiver Inclusion Criteria

  * Adult (≥18 years) relative or friend of a participating patient who the patient identifies as living with or has in-person contact with them at least twice per week.

Exclusion Criteria:

- Patient Exclusion Criteria

* Patients with a diagnosis of acute promyelocytic leukemia (APML)
* Patients with AML receiving supportive care alone
* Patients with psychiatric or cognitive conditions which the treating clinicians believe prohibits informed consent or compliance with study procedures
* Patients seen by a palliative care clinician (MD, DO, APP) during two previous hospitalizations in the six months prior to enrollment
* Patients expected to be discharged within 2 days

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Quality of Life (QOL) | Over 12 weeks
  Establish that primary palliative care is non-inferior to specialty palliative care in patient-reported quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leukemia) over 12 weeks.
  Higher scores on FACT-Leukemia (range 0-176) indicate a better QOL.

SECONDARY OUTCOMES:
Patient Quality of Life (QOL) | Up to 2 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with respect to patient-reported quality of life (QOL) as measured by the Functional Assessment of Cancer Therapy-Leukemia (FACT-Leukemia).
Patient Depression Symptoms | Up to 12 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with depression symptoms as measured by the Hospital Anxiety and Depression Scale (HADS).
  Higher scores on HADS depression subscale (range 0-21) indicate greater depression symptoms.
Patient Anxiety Symptoms | Up to 12 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with anxiety symptoms as measured by the Hospital Anxiety and Depression Scale (HADS).
  Higher scores on HADS anxiety subscale (range 0-21) indicate greater anxiety symptoms.
Patient Post-Traumatic Stress Disorder (PTSD) Symptoms | Up to 12 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with respect to post-traumatic stress (PTSD) symptoms as measured by the Post-Traumatic Stress Checklist-Civilian version.
  Higher scores on the Post-Traumatic Stress Checklist (range 17-85) indicate greater PTSD symptoms.
End-of-Life (EOL) Communication | Up to 12 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with respect to patient reported end-of-life (EOL) communication measured by the Prognostic Awareness Impact Scale (PAIS).
  The PAIS includes an item that measures patient self-report of communication about their wishes if they were dying (yes vs. no).
End-of-Life (EOL) Care | Last 30 days of life
  Assess whether primary palliative care is non-inferior to specialty palliative care with respect to chemotherapy administration in the last 30 days of life based on documentation from the Electronic Health Record.
Caregiver Quality of Life (QOL) | Up to 12 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with respect to caregiver quality of life measured by the Caregiver Oncology QOL Questionnaire (CARGOQOL).
  Higher scores on CARGOQOL (range 0-100) indicate better QOL.
Caregiver Burden | Up to 12 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with respect to caregiver burden measured by the Caregiver Reaction Assessment (CRA).
  Higher scores on the CRA (range 24-120) indicate greater caregiving burden.
Caregiver Depression Symptoms | Up to 12 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with respect to caregiver depression symptoms measured by the Hospital Anxiety and Depression Scale (HADS).
  Higher scores on HADS depression subscale (range 0-21) indicate greater depression symptoms.
Caregiver Anxiety Symptoms | Up to 12 Weeks
  Assess whether primary palliative care is non-inferior to specialty palliative care with respect to caregiver anxiety symptoms measured by the Hospital Anxiety and Depression Scale (HADS).
  Higher scores on HADS anxiety subscale (range 0-21) indicate greater anxiety symptoms.

OTHER OUTCOMES:
Patient Prognostic Understanding | Up to 24 weeks
  Compare patient prognostic understanding between those receiving primary palliative care and specialty palliative care based on the Prognostic Awareness Impact Scale (PAIS). The PAIS items that focus on the likelihood of cure will be used to compare prognostic understanding. Patients will report the likelihood of cure of their leukemia on a Likert's scale. Prognostic understanding will be dichotomized into likely cure versus. unlikely cure and compared between the two groups.
Patient Coping | Up to 24 weeks
  Compare patient coping between those receiving primary palliative care versus specialty palliative care using the Brief Cope. Higher scores on the domains of the Brief Cope indicate higher use of coping strategies.
Hospitalization | Last 30 days of life
  Compare hospitalization in the last 30 days of life between those receiving primary palliative care versus specialty palliative care.
Intensive Care Unit (ICU) Admissions | Last 30 days of life
  Compare intensive care unit admissions in the last 30 days of life between those receiving primary palliative care versus specialty palliative care.
Hospice Utilization | Last 30 days of life
  Compare hospice utilization between those receiving primary palliative care versus specialty palliative care.
Hospice Length of Stay | Last 30 days of life
  Compare hospice length of stay between those receiving primary palliative care versus specialty palliative care.
Patient Symptom Burden | Up to 24 weeks
  Compare patient symptom burden between those receiving primary palliative care versus specialty palliative care using the revised Edmonton Symptom Assessment Scale (ESAS-R).
  Higher scores on ESAS-R (range 0 - 100) indicate greater symptom burden.
Patient Perception of Care | Up to 24 weeks
  Compare patients' perception of patient-centeredness of care between those receiving primary palliative care versus specialty palliative care using the Patient Perception of Patient-Centeredness of Care (PPPC).
  Higher scores indicate greater satisfaction with care.
Caregiver-Reported End-of-Life (EOL) Communication | Up to 24 weeks
  Compare caregiver-reported end-of-life (EOL) communication between those receiving primary palliative care versus specialty palliative care measured by the Prognostic Awareness Impact Scale (PAIS). The PAIS includes an item that measures patient self-report of communication about their wishes if they were dying (yes vs. no).
Caregiver Prognostic Understanding | Up to 24 weeks
  Compare caregiver prognostic understanding between those receiving primary palliative care versus specialty palliative care based on the Prognositic Awareness Impact Scale (PAIS). PAIS items that focus on likelihood of cure will be used to compare prognostic understanding.
Caregiver Coping | Up to 24 weeks
  Compare caregiver coping between those receiving primary palliative care versus specialty palliative care using the Brief COPE. Higher scores on the domains of the Brief Cope indicate higher use of coping strategies.

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital; Jennifer Temel, MD, Principal Investigator — Massachusetts General Hospital
Locations (20):
- United States (20):
  - University of Alabama - Birmingham, Birmingham, Alabama
  - Stanford University, Stanford, California
  - University of Colorado Denver I Anschutz Medical Campus, Denver, Colorado
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Evanston, Illinois
  - Indiana University, Bloomington, Indiana
  - Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - University of Rochester, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University, Durham, North Carolina
  - Ohio State University, Columbus, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation